CLINICAL TRIAL: NCT04458025
Title: Prospective, Randomized Clinical Trial Comparing Early Versus Delayed Postoperative Mobilization After Arthroscopic Rotator Cuff Tear Reapair.
Acronym: RAPIDREHAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Borja Alcobía-Díaz MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Borja Alcobía-Díaz MD, PhD, MD, PhD, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAPIDREHAB
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Rotator Cuff Tear Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard rehabilitation program (Active Comparator): Standard postoperative 4 weeks immobilization rehabilitation program with a sling in adduction and internal rotation
  Interventions: Other: Standard rehabilitation program
- Early rehabilitation program (Experimental): Early rehabilitation program will start passive mobilization during second week after surgery, including controlled external rotation movements
  Interventions: Other: Early rehabilitation program

INTERVENTIONS:
Other: Standard rehabilitation program — Standard rehabilitation will start 4 weeks after surgery according to the standard of cre
  Arms: Standard rehabilitation program
Other: Early rehabilitation program — Early rehabilitation program will start 2 weeks
  Arms: Early rehabilitation program

SUMMARY:
Arthroscopic suture for complete and partial >50% thickness Rotator Cuff Tears (RCT) is the gold standard. However, there is no evidence of superiority of delayed postoperative mobilization protocols versus early ones, in terms of ROM, pain, quality of life and complications in last review published in 2019 by AAOS. Although, excessive immobilization can lead into stiffness, neuropathic pain or adhesive capsulitis. All of these are complications which can diminish patient quality of life or prolong their return to work or sports activities.

This is an experimental, prospective, non-blind, comparative, randomized clinical trial, between two options of treatment. On one treatment branch, we will continue applying our standard postoperative 4 weeks immobilization rehabilitation program with a sling in adduction and internal rotation. On the other treatment branch, we will start passive mobilization during second week after surgery, including controlled external rotation movements. All recruited patients will be followed-up during 12 months.

Our main objective is to compare differences in terms of functionality (using ASES scale). Secondary objectives are to compare differences in terms of ROM, functionality (using CMS and UCLA scales), pain (using VAS score), need of analgesic drugs, quality of life (using EQ-5D scale), return to previous work and sports activities, patient adhesion to protocol, complications and MRI rotator cuff retear ratio at 12 months follow-up.

After this study, we hope to develop a new postoperative mobilization protocol for patients. This protocol will be focused on timing, and self-administrated exercises in order to involve patients in their recovery, in the fastest and safest way for them.

ELIGIBILITY:
Inclusion Criteria:

* Age: Less tan 70 years old.
* Sex: Male or Female.
* Treatment: Arthroscopic RCT suture.
* RCT type: Degenerative, total or partial >50% thickness, less than 3 cm length tear.
* MRI Tear Classification: Patté's in coronal view I or II, Goutalier's <2, Fukuda's <2 and Seebauer´s 1A maximum.

Exclusion Criteria:

* Not meet the inclusion criteria.
* Previous surgical procedure in affected shoulder.
* Have been treated with 2 or more glucocorticoid injections in last year.
* High anesthetic risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Functionality | 12 months after surgery
  Functionality assessment using ASES scale

SECONDARY OUTCOMES:
Functionality-Constant-Murley scale | 12 months after surgery
  Functionality assessment using Constant-Murley scale
Functionality-UCLA | 12 months after surgery
  Functionality assessment using UCLA scale
Pain | 12 months after surgery
  Pain estimation according to visual analogic scale
Range of motion | 12 months after surgery
  Range of motion measured in degrees of a circle
Analgesic use | 12 months after surgery
  Need of analgesic drugs during the follow up period
Quality of life | 12 months after surgery
  Quality of life according to EQ-5D scale
Complications | 12 months after surgery
  Complications related to the surgery or rehabilitation
MRI rotator cuff retear ratio | 12 months after surgery
  MRI rotator cuff retear ratio determinate by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Borja Alcobía Díaz, MD PhD, Principal Investigator — Hospital Clinico San Carlos

IPD SHARING:
Plan to Share IPD: Undecided